CLINICAL TRIAL: NCT04663386
Title: Switch of Budesonide-formoterol Dry Powder Inhalers at Pharmacy in Norway; A Retrospective, Observational Study to Evaluate the Impact on Disease Control in Patients With Asthma and/or Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Switch of Budesonide-formoterol Dry Powder Inhalers at Pharmacy in Norway
Acronym: BufoSwitch
Status: Terminated | Type: Observational
Why Stopped: Target recruitment not reached
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 3103018
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Budesonide-Formoterol — Dry powder inhaler

SUMMARY:
This is a retrospective, multicentre, non-interventional, observational study in patients with asthma and/or COPD who are treated with budesonide-formoterol.

DETAILED DESCRIPTION:
In July 2018 Norwegian authorities decided to allow switch at pharmacy for dry powder inhalers (DPIs) containing budesonide-formoterol. Pharmacists are instructed to switch patients to the inhaler with the lowest price. The pharmacist will train the patient on how to use the new inhaler. All patients whose eligible inhaler switch occurred between 1st July 2018 and 1st March 2019 will be eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained.
2. Male or female patients with a diagnosis of asthma and/or COPD whose budesonide-formoterol DPI was switched to another budesonide-formoterol DPI at pharmacy between 1st July 2018 and 1st March 2019 (referred to as the eligible switch).
3. Age ≥12 years at time of switch.
4. Treated with budesonide-formoterol for at least 12 months before the eligible switch (pre-switch period) and 12 months after the eligible switch (post-switch period). Re-switch(es) of inhaler are allowed during the post-switch period.

Exclusion Criteria:

1. Patient has declined participation in the study or failed to respond to the invitation to participate.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with asthma and/or COPD treated with budesonide-formoterol DPI
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Disease control | 24 months
  The number of asthma and/or COPD exacerbations during the 12 months pre-switch and the 12 months post-switch.

SECONDARY OUTCOMES:
Budesonide-formoterol dose | 24 months
  The change in the treatment dose of budesonide-formoterol at the time of the eligible switch and at the end of the post-switch period (e.g. 12 months post-switch).
Training at pharmacy | 24 months
  The correlation between inhaler training given at pharmacy and exacerbations.
Healthcare utilisation | 24 months
  The number of asthma and/or COPD related hospitalisations, emergency room visits and visits to physicians 12 months pre-switch and 12 months post-switch.
Inhaler switch | 24 months
  The number of re-switches after the first 'eligible' switch and the reasons for that switch.

CONTACTS AND LOCATIONS:
Overall Officials: Jorn Ossum, Principal Investigator — Flattum Legesenter
Locations (1):
- Flattum Legesenter, Hønefoss, Norway

IPD SHARING:
Plan to Share IPD: No